CLINICAL TRIAL: NCT01308463
Title: Discovery Elbow Long-Term Survivorship Study
Brief Title: Discovery Elbow Long-Term Survivorship
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to change in sponsorship
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.EX002
Record Dates: First submitted 2010-07-23; First posted 2011-03-04 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Survivorship; Pain
Keywords: elbow long-term Survivorship; Study participant Discovery Elbow Multi-center Study who; consent for the Discovery Elbow Long-term SurvivorshipStudy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Discovery elbow minimally constrained — patient participating in the Discovery Elbow Multi-center study

SUMMARY:
The Discovery™ Elbow Multi-Center Prospective Study (5-year Study) patients will be consented at the two year or next scheduled follow-up period for the early-enrolled patients.

DETAILED DESCRIPTION:
Eligibility: Patient(s) must be enrolled in the Discovery Multi-Center Prospective Study. The patient must consent to participation in the Discovery Long-term Survivorship Study.

In order to continue to follow the multi-center subjects long-term Biomet would like to extend the follow-up to include annual follow-ups from 10 to 15 years to document long-term survivorship. The annual follow-up will be obtained by sending annual questionnaire directly to the patients by mail. The Patient ASES questionnaire and survivorship data questions will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in the Discovery Elbow Multi-center Study
2. Consent to participate in the Discovery Elbow Long-Term Survivorship Study

Exclusion Criteria:

1. Patient is not a Discovery Elbow Multi-center Participant
2. Patient does not provide consent for the Discovery Elbow Long-term Survivorship Study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Study population shall be participanting in the Discovery Elbow Multi-center Study who provide consent for the Discovey Elbow Long-term Survivoship Study
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, PhD, Study Director — Director Clinical Research, Biomet Orthopedics, LLC
Locations (4):
- United States (4):
  - Florida Orthopedic Institute, Tampa, Florida
  - The Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vanderbilt Hand Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment has been discontinued.
Groups:
- Discovery Elbow: This arm includes all subjects who underwent total elbow arthroplasty with the Discovery Total Elbow and entered the long-term survival study.
Period: Overall Study
Arm/Group | Discovery Elbow
Started | 29
6 Months | 23
1 Year | 21
2 Years | 18
3 Years | 17
4 Years | 20
5 Years | 20
6 Years | 11
7 Years | 12
8 Years | 14
9 Years | 11
10 Years | 8
11 Years | 8
12 Years | 2
Completed | 0
Not Completed | 29
Not completed — Study Discontinued | 23
Not completed — Death | 4
Not completed — Revision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Discovery Elbow
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
Hand Dominance [Count of Participants; unit: Participants]
  Ambidextrous | 1
  Left | 2
  Right | 25
  Unknown | 1
Primary Diagnosis [Count of Participants; unit: Participants]
  Functional Deformity | 1
  Humeral Fracture | 3
  Osteoarthritis | 2
  Other | 4
  Rheumatoid Arthritis | 11
  Traumatic Arthritis | 7
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Derived American Shoulder and Elbow Society (ASES) Pain Score
Description: This is the patient's perception of pain related to the operative elbow. Maximum pain score = 50 (worst) Minimum pain score = 0 (best)
Time Frame: 10 Years Post-op
Population: The number of participants analyzed in this section is reflective of the number of participants/elbows with the complete data required to calculate this score. This is different than the number reflected in participant flow which is indicative of the number of participants/elbows with any data during the given interval.
Measure: Median (Standard Deviation); unit: units on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery Elbow
Number analyzed (Participants) | 9
Number analyzed (Elbows) | 9
units on a scale | 5.3 (6.8)

2. Primary Outcome: Patient Derived American Shoulder and Elbow Society (ASES) Function
Description: This is the patient's perception of function. The maximum score is 36 and the minimum score is 0. The maximum score represents maximum function.
Time Frame: 10 Years Post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery Elbow
Number analyzed (Participants) | 9
Number analyzed (Elbows) | 9
units on a scale | 25.1 (8.8)

3. Primary Outcome: Patient Derived American Shoulder and Elbow Society (ASES) Satisfaction
Description: This is the patient's perception of satisfaction with the elbow replacement surgery.
  Maximum Score = 10 Minimum Score = 0 Maximum Score represents maximum satisfaction.
Time Frame: 10 Years Post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Elbows
Arm/Group | Discovery Elbow
Number analyzed (Participants) | 9
Number analyzed (Elbows) | 9
units on a scale | 9.2 (1.4)

4. Secondary Outcome: Survivorship Will be Measured by the Incidence of Revision or Removals
Description: The consented Patient will answer specific questions about their elbow replacement such as; if the elbow replacement has been removed
Time Frame: 10 years Post-op
Population: This analysis cannot be conducted due to the low number of cases available with 10 year data. There is not sufficient data to calculate survivorship. This study is being terminated since the product has been sold to another company.
Units Other Than Participants: Elbows
Arm/Group | Discovery Elbow
Number analyzed (Participants) | 0
Number analyzed (Elbows) | 0

ADVERSE EVENTS:
Arm/Group | Discovery Elbow
Serious Adverse Events (participants affected / at risk) | 10/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discovery Elbow (N=29)
Infection in Operative Joint (Infections and infestations) | 1 (7) — Chronic infection and treatment of elbow
Complex Laceration of Arm (Skin and subcutaneous tissue disorders) | 1 (1)
Ulnar Bearing Loosening (Surgical and medical procedures) | 1 (1) — bearing exchange
Screw Loose from Bearing (Surgical and medical procedures) | 1 (1) — Bearing revision
Bushing Failure (Surgical and medical procedures) | 1 (1) — Squeaking in elbow. X-rays show bushing failure.
Unspecified Events Leading to Death (General disorders) | 4 (4) — Death
TEA Revision (Surgical and medical procedures) | 1 (1)
Revision - Loose Humeral Component (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
The early termination of this study lead to only a small number of consenting subjects available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A publication which uses data in addition to the authors will be reviewed by all who have contributed data, and all of the contributors will be recognized.

All publications will be reviewed by BIOMET at least 30 days prior to publication.